CLINICAL TRIAL: NCT04490876
Title: Outcomes of Extensive Brilliant Blue G-Assisted Internal Limiting Membrane Peeling in Retinal Detachment With Proliferative Vitreoretinopathy Using 3D Visualization System
Brief Title: Outcomes of Extensive Brilliant Blue G-Assisted Internal Limiting Membrane Peeling in Proliferative Vitreoretinopathy
Acronym: ILM
Status: Completed | Type: Observational
Sponsor: Centro Oftalmológico Dr Charles (Other)
Responsible Party: Principal Investigator, Anibal Andres Francone, Medical Doctor. Ophthalmologist Board Certificate. Fellowship in Vitreoretinal Diseases., Centro Oftalmológico Dr Charles
Other Study IDs: 3701001
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: Retinal Detachment; Proliferative Vitreoretinopathy; Internal Limiting Membrane; ILM peeling; Brilliant Blue G
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinal Detachment with PVR: Proliferative vitreoretinopathy (PVR), a major complication of rhegmatogenous retinal detachment (RRD), is an abnormal process whereby proliferative, contractile cellular membranes form in the vitreous and on both sides of the retina, resulting in tractional retinal detachment with fixed retinal folds. Patients with RD complicated by PVR will be included, and the proposed intervention will be performed.
  Interventions: Procedure: 3D Pars Plana Vitrectomy associated with Extensive Brilliant Blue G-Assisted ILM Peeling Method

INTERVENTIONS:
Procedure: 3D Pars Plana Vitrectomy associated with Extensive Brilliant Blue G-Assisted ILM Peeling Method — After the injection of Brilliant Blue-G (BBG) into the vitreous cavity, the epiretinal membrane (ERM) with cellular proliferation on the surface of the retina did not stain clearly, while the internal limiting membranes did stain clearly. We peeled off the internal limiting membrane (ILM) underlying the ERM using the ILM forceps for the macular area and the serrated forceps for the remaining ILM beyond the vascular arcades (Grieshaber, Alcon Laboratories, Inc., Fort Worth, Texas (Figure1) and enhanced membrane viewing with filters on the Ngenuity system. Restaining with BBG was needed and perfluorocarbon liquid PFCL was injected with a coaxial Dual Bore cannula (MedOne) to flatten the retina.

SUMMARY:
The aim of this study is to report outcomes of pars plana vitrectomy (PPV) in retinal detachment (RD) accompanied with proliferative vitreoretinopathy (PVR) after extensive Brilliant Blue G-Assisted internal limiting membrane (ILM) peeling using a 3D visualization system.

This is retrospective consecutive case series of 14 eyes treated with PPV for RD repair. The patients were follow for 7 to 47 months (mean follow-up: 14.1 months ).

DETAILED DESCRIPTION:
This is the retrospective study of 14 consecutive patients suffering from retinal detachment with proliferative vitreoretinopathy who underwent primary PPV at the Department of Retina of Centro Oftalmologico Dr Charles, Buenos Aires-Argentina between January 1, 2016 and August 1, 2020 . This study followed the tenets of the Declaration of Helsinki and it was approved by the approved by the research ethics committee (www.comitedeeticaceic.com.ar). Written informed consent was taken from all subjects. All cases were performed by a single experienced vitreoretinal surgeon (MCH)

The treatment chosen in the study was pars plana vitrectomy with Brilliant Blue G (BBG) staining using the Ngenuity 3D Visualization System (Alcon). We spread 0.05% w/v BBG solution (OCUBLUE PLUS, Aurolab), approximately 0.3-0.5 ml, on the retinal surface and peeled off the ILM from the posterior pole up to the periphery, thus ensuring the total removal of the overlying epiretinal membranes responsible for recurrent detachment. Frequent restaining with BBG helped revealing new edges and perfluorocarbon liquid was used in others to stabilize the retina (Figure1). ).. All patients underwent vitreoretinal surgery due to RD (rhegmatogenous, tractional or combined rhegmatogenous and tractional). Exclusion criteria from the study was the time of follow-up less than 6 months.

Average age at the time of the presence of RD was 56 ± 8.7 years (range 23-77 years). Pre- and postoperative data were collected. Descriptive statistical analysis included gender, age at the presentation, laterality, etiology, duration of presenting symptoms, presences of ocular comorbidities, macular status (attached or non-attached), presence of PVR (preretinal, subretinal and intraretinal) initial and final best-corrected visual acuity (BCVA), number of procedures, type of endotamponade during PPV, final lens status, duration of the follow-up, anatomical success and complications. Indications for PPV were as follows: presence of advanced PVR and/or total RD and/or multiple breaks, giant retinal tears. PVR was graded according to the Retina Society Terminology Classification and anatomical location (references). Visual acuity was measured by Snellen charts. The anatomical success was defined as persistent retinal reattachment at the last follow-up visit (in absence of silicone oil tamponade).

Statistical computations were performed using STATA 16 data analysis and statistical software (StataCorp LLC, College Station, Texas, USA)

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years age suffering from retinal detachment with proliferative vitreoretinopathy who underwent primary PPV at the Department of Retina of Centro Oftalmologico Dr Charles, Buenos Aires-Argentina between January 1, 2016 and August 1, 2020 .

Exclusion Criteria:

* patients younger than 18 years age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private retina clinic.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Persistent retinal reattachment | 6 months after silicone oil removal
  The anatomical success was defined as persistent retinal reattachment at the last follow-up visit (in absence of silicone oil tamponade).

SECONDARY OUTCOMES:
Mean Best Corrected Visual Acuity | mean follow-up: 14.1 months
  BCVA was recorded at each visit, reported in Snellen fraction and converted into logarithm of the minimal angle of resolution (logMAR) values for statistical analysis.
Spectral Domain OPTICAL COHERENCE TOMOGRAPHY (SD-OCT) IMAGING of the MACULA | mean follow-up: 14.1 months
  SD-OCT images were obtained with the Spectralis OCT with eye-tracking dual-beam technology (Heidelberg Engineering GmbH, Heidelberg, Germany) and reviewed with the Heidelberg Eye Explorer (version 1.8.6.0) using the HRA/Spectralis Viewing Module (version 5.8.3.0). All patients underwent the Sequential 12-line radial scans and were evaluated for the presence of intraretinal/subretinal fluid. Mean central foveal thickness was obtained with the automated ''thickness map'' function of the Heidelberg Eye Explorer.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Oftalmologico Dr Charles, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Foveau P, Leroy B, Berrod JP, Conart JB. Internal Limiting Membrane Peeling in Macula-off Retinal Detachment Complicated by Grade B Proliferative Vitreoretinopathy. Am J Ophthalmol. 2018 Jul;191:1-6. doi: 10.1016/j.ajo.2018.03.037. Epub 2018 Apr 3. PMID 29621507
- [Result] Odrobina DC, Michalewska Z, Michalewski J, Nawrocki J. High-speed, high-resolution spectral optical coherence tomography in patients after vitrectomy with internal limiting membrane peeling for proliferative vitreoretinopathy retinal detachment. Retina. 2010 Jun;30(6):881-6. doi: 10.1097/IAE.0b013e3181c96952. PMID 20182404
- [Result] Sakamoto H, Yamanaka I, Kubota T, Ishibashi T. Indocyanine green-assisted peeling of the epiretinal membrane in proliferative vitreoretinopathy. Graefes Arch Clin Exp Ophthalmol. 2003 Mar;241(3):204-7. doi: 10.1007/s00417-002-0601-9. Epub 2003 Feb 20. PMID 12644944
- [Result] Aras C, Arici C, Akar S, Muftuoglu G, Yolar M, Arvas S, Baserer T, Koyluoglu N. Peeling of internal limiting membrane during vitrectomy for complicated retinal detachment prevents epimacular membrane formation. Graefes Arch Clin Exp Ophthalmol. 2009 May;247(5):619-23. doi: 10.1007/s00417-008-1025-y. Epub 2008 Dec 24. PMID 19107502
- [Result] Enaida H, Hisatomi T, Hata Y, Ueno A, Goto Y, Yamada T, Kubota T, Ishibashi T. Brilliant blue G selectively stains the internal limiting membrane/brilliant blue G-assisted membrane peeling. Retina. 2006 Jul-Aug;26(6):631-6. doi: 10.1097/01.iae.0000236469.71443.aa. PMID 16829804
- [Result] Kumar A, Hasan N, Kakkar P, Mutha V, Karthikeya R, Sundar D, Ravani R. Comparison of clinical outcomes between "heads-up" 3D viewing system and conventional microscope in macular hole surgeries: A pilot study. Indian J Ophthalmol. 2018 Dec;66(12):1816-1819. doi: 10.4103/ijo.IJO_59_18. PMID 30451186
- [Result] Lai CT, Kung WH, Lin CJ, Chen HS, Bair H, Lin JM, Chen WL, Tien PT, Tsai YY. Outcome of primary rhegmatogenous retinal detachment using microincision vitrectomy and sutureless wide-angle viewing systems. BMC Ophthalmol. 2019 Nov 19;19(1):230. doi: 10.1186/s12886-019-1238-3. PMID 31744475